CLINICAL TRIAL: NCT01975038
Title: Adaption of the Skin Sun Sensitivity Scale for People With All Pigment Varieties
Brief Title: Adaption of the Skin Sun Sensitivity Scale
Status: Completed | Type: Observational
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, June Robinson, Research Professor of Dermatology (MD), Northwestern University
Other Study IDs: STU00086547
Record Dates: First submitted 2013-10-28; First posted 2013-11-04 (Estimated); Last update posted 2014-08-01 (Estimated); Status verified 2014-07

CONDITIONS: Skin Diseases
Keywords: Melanin Index; Fitzpatrick Skin Phototype; Spectrophotometry; Skin Diseases
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A convenience sample: The characteristics of the sample will be monitored to assure that each category of skin type (I- VI) is accrued in sufficient size to support analysis. In addition, the sample will have equal representation from 4 ethnic groups within each skin type category: African American, Asian, Hispanic, or non-Hispanic White. Participants will self-identify as being Asian, Black, Hispanic Black, Hispanic White, or non-Hispanic White.

SUMMARY:
Determining Fitzpatrick skin phototypes (FST) allows physicians to assess a person's risk of developing sunburn, and thus the need for sun protection to prevent the development of skin cancer. Reflectance spectrophotometry objectively measures the melanin index (MI) and can assist in determining the accuracy of self-reported FST compared with dermatologist-determined FST. At present, we seek to determine the accuracy of an adapted Skin Sun Sensitivity Scale for individuals of all pigmentation varieties (FST I through VI) as compared with spectrophotometric measurements assessing FST. Our principal objective is to correlate the MI under usual conditions by spectrophotometry with the adapted Fitzpatrick SPT as determined by the patients' responses to the adapted questionnaire.

DETAILED DESCRIPTION:
1. BACKGROUND AND RATIONALE:

   We extended the pilot study (IRB STU27549) of our objective measurement of skin pigmentation with correlation to the self-reported skin reaction to sun exposure to a larger sample with special emphasis on people with skin of color and compare the results to those obtained by spectrophotometry. We found that forty-two percent (114 of 270) of the participants' responses to the burning and tanning questions could not be classified using standard Fitzpatrick skin phototype (FST) definitions. At present, we seek to determine the accuracy of an adapted Skin Sun Sensitivity Scale for individuals of all pigmentation varieties (FST I through VI) as compared with spectrophotometric measurements assessing FST.

   Fitzpatrick Skin Phototyping Skin phototyping has usually been determined subjectively by trained investigators or clinicians using sun burning and/or sun tanning responses. In addition, subject self-report of ease of sunburning and tanning is used in surveys to determine the risk of developing skin cancer. (Table 1) Responses to the Fitzpatrick Skin Phototype (SPT) questions may be unreliable due to recall bias, subjective bias by clinicians and subjects, lack of cultural sensitivity of the questions, and the subjects' use of sun protection behaviors from early childhood such that the subject may not have experienced sunburn.

   Table 1. Skin type; Erythema and Tanning Reactions to the First Summer Exposure I Always burns, never tan (painful burn at 24 hrs and no tan at 7d) II Burn easy, then develop light tan (painful burn at 24 hrs and a light tan at 7d) III Burn moderately, then develop light tan (slightly tender burn at 24 hrs, moderate tan at 7d) IV Burn minimally-rarely, then develop moderate tan (no burn at 24 hrs and a good tan at 7d) V Never burns, always develops dark tan VI Never burns, no noticeable change in appearance

   Unreliable Sunburning History A limitation of the 6 integer Roman numeral Fitzpatrick SPT was reliance upon a history of sunburn after the first exposure of the summer. For those who reside in regions that have sun exposure all year (e.g. Arizona, Florida, California), the sunburning-tanning question after the first exposure of the summer was often irrelevant. Lastly, in the 1990s people began to use sunscreens to prevent sunburns, thus, those with sun sensitive skin may never have experienced sunburn and were unable to answer the question about ease of sun burning.

   Multi-ethnic Populations There has been a tendency to group all people of a similar ethnic group into a single category of SPT, which introduces potential bias into the subjective assessment of SPT by investigators. For example, Hispanic whites are often considered "brown" and assigned to Skin Type IV (Table 2). The heterogeneity of those with multi-ethnic backgrounds makes it difficult to assess susceptibility to skin cancer on the basis of skin color, which is predominantly determined by pigments such as hemoglobin, melanin, bilirubin, and carotene.

   Skin Phototyping by Sunburning Ability. Skin Phototype Appearance Sunburning ability I Very white or freckled Always burn II White Usually burn III White to Olive Sometimes burn IV Brown Rarely burn V Dark brown Very rarely burn VI Black Never burn

   Over the last 3 decades, the Fitzpatrick SPT evolved from its original purpose of determining the amount of ultraviolet light (UVL) for treatment of psoriasis patients living in New England to become an assessment tool for skin cancer risk. As part of this evolution, the original 4 skin types (I-IV), that assessed sun reactivity with standardized questions about the ease of sun burning and tanning reactions to the first summer sun exposure, were modified by adding SPT V and VI to include those with brown and black skin.

   Our research demonstrated that the SPT modifications to include people with skin of color were neither culturally sensitive nor accurate as people of color were unable to respond to the questions about their experience with sunburn and tanning. People with skin of color did not report becoming red or pink but rather experienced "irritation" after sun exposure. In our recently reported work, we proposed a modification of the FST questions to allow people with skin of color to be able to respond (Survey questions 1and 2). We now wish to test the responses of people to these self-report questions and compare the responses with the melanin index as determined by spectrophotometry.(Survey question 9)

   Spectrophotometry The "gold standard" method of assessing skin pigmentation is reflectance spectrophotometry (RS). Pershing et al performed seminal research comparing the area under the curve obtained by RS to profile the constitutive skin color with clinicians' assessment of SPT. For skin types I-III, Pershing et al (2008) found inconsistency between clinicians' and reflectance spectrophotometric (RS) assessments of SPT. The clinicians adjusted the patients' SPT as determined by their historical sun burning and tanning response by factoring in observed hair and eye color. For example, red-haired individuals determined by RS to be SPT III were listed as SPT I by clinical dermatologists. Subjective assessment of SPT by clinicians was heavily influenced by patients' hair and eye color. The Pershing study, which accrued 125 subjects did not accrue sufficient numbers of subjects with skin of color (Skin types III-VI) to be able to report meaningful results. (I 20; II 53, III 21, IV 10, V 16, VI 5)

   It should be noted that the area under the curve obtained by RS includes the red reflectance, thus, it is does not solely represent skin pigmentation. Skin pigmentation or melanin provides photoprotection and can be calculated as melanin index, MI. (see following section on Melanin Index) Even as early as 1961, the potential for confounding of the MI obtained by RS by dilatation of superficial blood vessels was recognized. The device, Mexameter MX 18, internally corrects for the red reflectance in calculating the melanin index. The melanin index is derived from the multilayered skin model and Lambert-Beer's law.

   Significance:

   While those that are at risk to develop skin cancer have less melanin content (skin type I) than those at low risk (skin type VI), people with skin phototypes in the mid-range (III and IV) believe that their natural skin tone is protective against sunburns, thus, they fail to use sun protection. When people with skin type III and IV are exposed to more intense ultraviolet light in more southern latitudes than Chicago they are surprised by the sunburn they experience. In our proof of principle research, people with skin type III and IV, who viewed the image of their skin on the computer screen, perceived that the "color was grainy" and made the conclusion that the "holes" in their skin pigment made it possible for them to burn

   This study will further objectively measure the MI of people with skin of color. Thus, it is essential that we accrue a representative sample of people with skin of color with all ethnic groups represented over the greatest range of skin types for those self-identifying themselves as members of the group.
2. STUDY OBJECTIVES:

Our principal objective is to correlate the melanin index under usual conditions by spectrophotometry with the adapted Fitzpatrick SPT as determined by the patients' responses to the adapted questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Are at least 18 years old
* Are fluent in English
* Are able to complete the study procedures including answering questionnaires
* Are willing to have spectrophotometry readings taken of right upper inner arm

Exclusion Criteria:

* Used self-tanning products or tan accelerators on the right upper inner arm in the 4 weeks prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A convenience sample of approximately 200 Northwestern University students, employees (faculty and staff), patients attending the dermatology clinic, and attendees of Northwestern University dermatology-related events will be selected for measurement of the melanin index with the Mexameter MX18.
  The characteristics of the sample will be monitored to assure that each category of skin type (I- VI) is accrued in sufficient size to support analysis. In addition, the sample will have equal representation from 4 ethnic groups within each skin type category: African American, Asian, Hispanic, or non-Hispanic White. Participants will self-identify as being Asian, Black, Hispanic Black, Hispanic White, or non-Hispanic White.
Sampling Method: Non-Probability Sample
Enrollment: 292 (Actual)
Dates: Start 2013-10; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Melanin Index by Spectrophotometry | At baseline
  Spectrophotometer measurement is the wavelength of the reflected light measured in nm. It represents the area under the curve for the all wavelengths of light, thus a reading will be expressed as (192 ±30, mean ± SD).

SECONDARY OUTCOMES:
Participant Self-Report of Fitzpatrick Skin Type | At baseline
  Subjects will be asked to respond to the standard survey questions about ease of sunburning and tanning. (Q1, 2)
Assessment of Ease of Freckling as a Child and Ethnicity | At baseline
  Subjects will be asked to respond to standard questions self-reporting ease of freckling as child of about 10 years old and ethnic background. (Q3,4,7)
Assessment of Fitzpatrick Skin Type using the Adapted Skin Phototype Measure | At baseline
  Trained personnel will review interview the subjects' response to survey items 1 and 2 and assign a SPT determined by their responses. (Q9)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis P West, PhD, Study Director — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

REFERENCES:
- [Background] Chan JL, Ehrlich A, Lawrence RC, Moshell AN, Turner ML, Kimball AB. Assessing the role of race in quantitative measures of skin pigmentation and clinical assessments of photosensitivity. J Am Acad Dermatol. 2005 Apr;52(4):609-15. doi: 10.1016/j.jaad.2004.03.051. PMID 15793510
- [Background] Chung JH, Koh WS, Youn JI. Relevance of skin phototyping to a Korean population. Clin Exp Dermatol. 1994 Nov;19(6):476-8. doi: 10.1111/j.1365-2230.1994.tb01250.x. PMID 7889667
- [Background] Dawson JB, Barker DJ, Ellis DJ, Grassam E, Cotterill JA, Fisher GW, Feather JW. A theoretical and experimental study of light absorption and scattering by in vivo skin. Phys Med Biol. 1980 Jul;25(4):695-709. doi: 10.1088/0031-9155/25/4/008. PMID 7454759
- [Background] Diffey BL, Oliver RJ, Farr PM. A portable instrument for quantifying erythema induced by ultraviolet radiation. Br J Dermatol. 1984 Dec;111(6):663-72. doi: 10.1111/j.1365-2133.1984.tb14149.x. PMID 6508999
- [Background] Eilers S, Bach DQ, Gaber R, Blatt H, Guevara Y, Nitsche K, Kundu RV, Robinson JK. Accuracy of self-report in assessing Fitzpatrick skin phototypes I through VI. JAMA Dermatol. 2013 Nov;149(11):1289-94. doi: 10.1001/jamadermatol.2013.6101. PMID 24048361
- [Background] Feather JW, Ellis DJ, Leslie G. A portable reflectometer for the rapid quantification of cutaneous haemoglobin and melanin. Phys Med Biol. 1988 Jun;33(6):711-22. doi: 10.1088/0031-9155/33/6/005. PMID 3406055
- [Background] Fitzpatrick TB: Soleil et peau. J Med Esthet 1975, 2:33-34
- [Background] Fitzpatrick TB. The validity and practicality of sun-reactive skin types I through VI. Arch Dermatol. 1988 Jun;124(6):869-71. doi: 10.1001/archderm.124.6.869. No abstract available. PMID 3377516
- [Background] Kim M, Boone SL, West DP, Rademaker AW, Liu D, Kundu RV. Perception of skin cancer risk by those with ethnic skin. Arch Dermatol. 2009 Feb;145(2):207-8. doi: 10.1001/archdermatol.2008.566. No abstract available. PMID 19221276
- [Background] Lee JH, Kim TY. Relationship between constitutive skin color and ultraviolet light sensitivity in Koreans. Photodermatol Photoimmunol Photomed. 1999 Dec;15(6):231-5. doi: 10.1111/j.1600-0781.1999.tb00095.x. PMID 10599973
- [Background] Matts PJ, Dykes PJ, Marks R. The distribution of melanin in skin determined in vivo. Br J Dermatol. 2007 Apr;156(4):620-8. doi: 10.1111/j.1365-2133.2006.07706.x. PMID 17493065
- [Background] Melski JW, Tanenbaum L, Parrish JA, Fitzpatrick TB, Bleich HL. Oral methoxsalen photochemotherapy for the treatment of psoriasis: a cooperative clinical trial. J Invest Dermatol. 1977 Jun;68(6):328-35. doi: 10.1111/1523-1747.ep12496022. PMID 864273
- [Background] MONASH S. Skin color. A correlation of reflectance measurement and clinical appearance. Arch Dermatol. 1961 Oct;84:654-9. doi: 10.1001/archderm.1961.01580160118023. No abstract available. PMID 14475328
- [Background] National Institutes of Health. Strategic Research Plan to Reduce and Ultimately Eliminate Health Disparities Volume 1. Years 2002-2006 U.S. Department of Health and Human Services 2002.
- [Background] Park SB, Suh DH, Youn JI. Reliability of self-assessment in determining skin phototype for Korean brown skin. Photodermatol Photoimmunol Photomed. 1998 Oct-Dec;14(5-6):160-3. doi: 10.1111/j.1600-0781.1998.tb00035.x. PMID 9826886
- [Background] Pershing LK, Tirumala VP, Nelson JL, Corlett JL, Lin AG, Meyer LJ, Leachman SA. Reflectance spectrophotometer: the dermatologists' sphygmomanometer for skin phototyping? J Invest Dermatol. 2008 Jul;128(7):1633-40. doi: 10.1038/sj.jid.5701238. Epub 2008 Jan 17. PMID 18200057
- [Background] Robinson JK, Joshi KM, Ortiz S, Kundu RV. Melanoma knowledge, perception, and awareness in ethnic minorities in Chicago: recommendations regarding education. Psychooncology. 2011 Mar;20(3):313-20. doi: 10.1002/pon.1736. PMID 20878831
- [Background] Rubegni P, Cevenini G, Flori ML, Fimiani M, Stanghellini E, Molinu A, Barbini P, Andreassi L. Relationship between skin color and sun exposure history: a statistical classification approach. Photochem Photobiol. 1997 Feb;65(2):347-51. doi: 10.1111/j.1751-1097.1997.tb08569.x. PMID 9066310
- [Background] Shono S, Imura M, Ota M, Ono S, Toda K. The relationship of skin color, UVB-induced erythema, and melanogenesis. J Invest Dermatol. 1985 Apr;84(4):265-7. doi: 10.1111/1523-1747.ep12265342. PMID 3981038
- [Background] Stanford DG, Georgouras KE, Sullivan EA, Greenoak GE. Skin phototyping in Asian Australians. Australas J Dermatol. 1996 May;37 Suppl 1:S36-8. doi: 10.1111/j.1440-0960.1996.tb01078.x. PMID 8713010
- [Background] Stern RS, Momtaz K. Skin typing for assessment of skin cancer risk and acute response to UV-B and oral methoxsalen photochemotherapy. Arch Dermatol. 1984 Jul;120(7):869-73. PMID 6732259
- [Background] Takiwaki H, Shirai S, Kanno Y, Watanabe Y, Arase S. Quantification of erythema and pigmentation using a videomicroscope and a computer. Br J Dermatol. 1994 Jul;131(1):85-92. doi: 10.1111/j.1365-2133.1994.tb08462.x. PMID 8043425